CLINICAL TRIAL: NCT02296450
Title: Quality of Life (QoL) Assessment in Cancer Patients and Survivors With Dermatologic Conditions Using Dermatologic QoL Instruments
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: 14-236
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Dermatologic Conditions
Keywords: Quality of Life (QoL); Assessment; 14-236; Patients and Survivors
MeSH Terms: conditions — Neoplasms | interventions — Quality of Life; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Quality of Life (QoL) Assessment: Patients involved in this study will have a wide range of dermatologic conditions for which they will be assessed and managed by the treating physician. An appropriate QoL instrument will be administered at the initial visit, and if applicable, at subsequent follow-up visit(s). Treatment of the dermatologic condition will be at physician's discretion based on the patient's presenting symptoms and is not an intervention itself within this study.
  Interventions: Behavioral: Quality of Life (QoL) Assessment

INTERVENTIONS:
Behavioral: Quality of Life (QoL) Assessment — Per physician's discretion, the patient (or, if applicable, patient's family member/ spouse/ caregiver for FDLQI) will complete one or more of the following dermatology-specific QoL instruments: Skindex-16, Skindex-29 DLQI (Dermatology Life Quality Index), FDLQI (Family DLQI) - for patient's family member/spouse/caregiver ONLY, CDLQI (Children's DLQI;Cartoon version) - for patient's under the age of 18 ONLY-written, CDLQI (Children's DLQI; Cartoon version) - for patients under the age of 18 ONLY - cartoon version, FACT-G (Functional Assessment of Cancer Thearpy-General), FACT-Melanoma (Functional Assessment of Cancer Therapy-Melanoma), SCI (Skin Cancer Index) FACT-EGFRI-18 (Functional Assessment of Cancer Therapy-Epidermal Growth Factor Receptor Inhibitor-18), HFS-14 (Hand-Foot Syndrome) OMWQ (Oral Mucositis Weekly Questionnaire), ESTEEM, Hairdex , Skindex-29 modified for hair loss, Itchy QoL,CADS (Chemotherapy-induced alopecia distress scale)
  Other Names: MELASQOL (Melasma QoL Questionnaire), MQ (Madarosis Questionnaire), CHIMES (The Children's International Muscositis Evaluation Scale), SDM-Q-9, WoSSAC, VF - 14, VFQ-25; Scalpdex, Face-Q Skin Cancer, PRO-CTCAE Cutaneous IP, Traditional Decisional Conflict Scale; ONYCHO (Nail-specific QoL questionnaire); FACT Lym (Functional Assessment of Cancer Therapy Lymphoma)

SUMMARY:
The purpose of this study is to see how skin conditions that are related to different kinds of cancer or cancer treatments affect a patient's overall well-being. Skin conditions are common in cancer patients and survivors. Sometimes, the skin condition is directly related to the cancer. Other times, these conditions are a side effect of cancer treatment. Patients in the study will be asked to fill out at least one questionnaire about how they feel about their skin condition. If the patient needs to be treated for their skin condition, they will be asked to complete the same questionnaire when they return for a follow-up visit. The investigators hope the study will improve our understanding of how cancer patients feel about their skin conditions. They also hope this study helps them learn how to improve the way we treat skin conditions in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients and survivors with a pre-existing dermatologic condition related to their underlying disease or completed/ongoing therapy for cancer, who present for assessment/management of their skin condition.
* Male or female patients at least 3 years and older
* NOTE: Informed Consent guidelines will be followed for minors
* First grade adult family members, spouses, and caregivers of patients with a Grade 2 or 3 or higher dermatologic condition related to their primary cancer or cancer treatment able to provide written informed consent

Exclusion Criteria:

* Cognitive or psychiatric deficit resulting in an inability to provide written informed consent

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients and survivors who present to MSKCC's Dermatology clinics in Manhattan, Basking Ridge, Haupaugge or West Harrison may be approached to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Estimated)
Dates: Start 2014-11-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) questionnaire | 5 years
  in cancer patients and survivors with dermatologic conditions. This is a nontherapeutic and nondiagnostic protocol to obtain quality of life assessments from cancer patients and survivors who have dermatologic conditions, whether related to cancer therapies, or directly related to the primary cancer diagnosis. Data will be collected by using one or more dermatology-specific QoL instruments based on the underlying skin condition/s.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Suffolk- Hauppauge, Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/